CLINICAL TRIAL: NCT05201313
Title: Randomised Controlled Trial to Evaluate the Efficacy of Local Anaesthetic Application in Spray for the Repair of 1st- 2nd Perineal Lacerations Following Vaginal Delivery
Brief Title: Efficacy and Safety of the Application of Local Anaesthetic in Spray to Repair of 1st- 2nd Perineal Lacerations
Acronym: LISPRAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Stefano Restaino, Principal Investigator, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0042698/P/GEN/ARCS
Record Dates: First submitted 2022-01-04; First posted 2022-01-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Vaginal Discharge; Perineum; Rupture; Analgesia
Keywords: perineal laceration; suturing; anesthetic
MeSH Terms: conditions — Vaginal Discharge; Rupture; Agnosia | interventions — Lidocaine; Mepivacaine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) of superiority, with two parallel treatment arms.
  Phase 3 study. Randomized controlled single-center perspective study.
Masking Description: Open label: due to the different methods of administration, the blindness of the obstetrician-gynecological team cannot be guaranteed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine spray (Experimental): nebulization 3 puffs of 10 mL Lidocaine hydrochloride 10% spray at a distance of 4-5 cm
  Interventions: Drug: Lidocaine Hydrochloride
- mepivacaine infiltration (Active Comparator): subcutaneous / submucosal infiltration depending on the type of perineal tear of 10 ml of 1% mepivacaine hydrochloride
  Interventions: Drug: Mepivacaine Injection

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — nebulization of 3 puffs of 10 mL Lidocaine hydrochloride 10% spray at a distance of 4-5 cm
  Other Names: ECOCAIN
  Arms: lidocaine spray
Drug: Mepivacaine Injection — subcutaneous / submucosal infiltration depending on the type of perineal tear of 10 ml of 1% mepivacaine hydrochloride
  Other Names: MEPIVACAINA CLORIDRATO
  Arms: mepivacaine infiltration

SUMMARY:
Randomized controlled trial aimed at evaluating the efficacy and safety of the use of a local anesthetic spray, commonly used in clinical practice as off-label, during the suturing of perineal lacerations in post-partum, comparing it with the standard technique that involves the infiltration of lacerated tissues, by administering a NRS card at the end of the procedure.

DETAILED DESCRIPTION:
The study aims to compare the effectiveness of pain treatment during the suturing of postpartum perineal lacerations with lidocaine spray vs skin infiltration. The hypothesis of the study is that the treatment of perineal pain with nebulization demonstrates comparable efficacy vs the infiltration of mepivacaine hydrochloride in a population of patients subjected to suturing of postpartum lacerations. Eligible women will be randomly assigned to receive, after wound disinfection and cleansing of bleeding with mild haemostasis:

1. nebulization 3 puffs of 10 mL Lidocaine hydrochloride 10% spray at a distance of 4-5 cm (experimental group).
2. subcutaneous / submucosal infiltration depending on the type of perineal laceration of 10 ml of 1% mepivacaine hydrochloride (control group).

Since there are no previous published studies, regarding the use of nebulized lidocaine hydrochloride for the suturing of perineal lacerations, the number of puffs chosen was chosen based on what is indicated on the technical data sheet of lidocaine hydrochloride and making use of previous studies in the gynecological field, but with other indications.

The suture will be made once anesthetic efficacy is achieved, as per pharmacological indications. The administration of the anesthetic and the suturing of the lacerations will be performed by the gynecologist or by the gynecology resident who will be working at that time in the delivery room, as is routinely done in our Clinic. The patients will be enrolled consecutively following the order generated by the randomization list itself. By filling in specific pre-set cards, the data will be collected.

Initially, the primary outcome was NRS at the beginning of suturing and NRS at the end of the procedure. In a second moment, the investigators thought it would be better to ensure that adequate analgesia (NRS<4) was achieved for all patients during suturing, rather than varying the dosage of the anesthetic itself. The investigators then decided to reassess pain at successive time points, evaluating it at 0, 2, 4, 12, and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* have a 1st or 2nd degree postpartum perineal laceration requiring suturing;
* have reached 37 gestational weeks;
* are over 18 years of age;
* had a top birth;
* are able to understand the Italian language;
* have a consent to participate in the study;

Exclusion Criteria:

- have received epidural anesthesia within 2 hours prior to delivery;

* had an operative birth;
* have a psychiatric pathology;
* have had a twin birth;
* have experienced adverse reactions to any local anesthetic in the past;
* hypersensitivity to the active substance or to any of the excipients
* Severe disturbances of the cardiac conduction system
* Acute non compensated heart failure
* Severe arteriopathies
* Severe uncontrolled hypertension
* Intravascular injections
* Septicemia Dysfunction
* Infection at the injection site
* Kidney failure. Providing for the exclusion of patients with severe renal impairment (estimated GFR <30 mL / min / 1.73 m2 at the time of screening).
* Advanced liver dysfunction
* Hyperthyroidism
* Acute angle glaucoma
* Participation in a clinical trial in which an investigational drug was administered within 30 days of screening or 5 half-lives of the study drug
* Any clinical condition that in the investigator's judgment would render the patient unsuitable for the study including, but not limited to, infectious, inflammatory, psychiatric, neurological, cardiological, renal, hepatic, respiratory, diabetes) conditions or laboratory value at clinically meaningful screening that, an investigator's opinion, may present a safety risk, interface with study compliance and follow-up;
* have had in pregnancy liver disease including pre-eclampsia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
NRS 2 | At 2 hours after delivery
  numeric rating scale for pain (0=no pain-10=maximum pain)
NRS 4 | At 4 hours after delivery
  numeric rating scale for pain (0=no pain-10=maximum pain)
NRS 12 | At 12 hours after delivery
  numeric rating scale for pain (0=no pain-10=maximum pain)
NRS 24 | At 24 hours after delivery
  numeric rating scale for pain (0=no pain-10=maximum pain)
NRS o | during suturing
  numeric rating scale for pain (0=no pain-10=maximum pain)

SECONDARY OUTCOMES:
need for additional doses (number of additional nebulizations, presence or absence of additional infiltration) | during the suture
  need for an additional dose of nebulization and / or additional infiltration during the suturing of the postpartum perineal laceration
final satisfaction, assessed via telephonic interview | 30 days follow up
  satisfaction of the puerpera, assessed through the 30 days-follow up, asking for the patient's opinion regarding postpartum pain and any long-term complications

CONTACTS AND LOCATIONS:
Overall Officials: Lorenza Driul, professor, Study Chair — DAME
Locations (1):
- ASUFC, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Restaino S, Degano M, Rizzante E, Battello G, Paparcura F, Biasioli A, Arcieri M, Filip G, Vetrugno L, Dogareschi T, Bove T, Petrillo M, Capobianco G, Vizzielli G, Driul L; LISPRAY Group. Lidocaine spray vs mepivacaine local infiltration for suturing 1st/2nd grade perineal lacerations: a randomised controlled non-inferiority trial. BMC Pregnancy Childbirth. 2024 Jun 24;24(1):439. doi: 10.1186/s12884-024-06640-7. PMID 38914976